CLINICAL TRIAL: NCT01490684
Title: Invasive Candidiasis in Critically Ill Patients in Saudi Arabia: A Prospective Cohort Study
Brief Title: Invasive Candidiasis in Saudi ICUs
Acronym: ICIP-SA
Status: Completed | Type: Observational
Sponsor: Hasan Al-Dorzi (Other Government)
Collaborators: King Fahad Medical City (Other Government)
Responsible Party: Sponsor-Investigator, Hasan Al-Dorzi, Consultant, Intensive Care Department, King Abdulaziz Medical City
Organization: King Abdulaziz Medical City (Other Government)
Other Study IDs: KAMC
Record Dates: First submitted 2011-12-02; First posted 2011-12-13 (Estimated); Results first posted 2018-08-24 (Actual); Last update posted 2018-08-24 (Actual); Status verified 2017-11

CONDITIONS: Invasive Candidiasis
Keywords: candidiasis; critically ill; outcomes
MeSH Terms: conditions — Candidiasis, Invasive; Candidiasis; Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Epidemiology and clinical outcomes of invasive candidiasis in critically ill patients in Saudi Arabia is not well studied. This observational study objectives include to determine the epidemiology, risk factors and outcomes of invasive Candida infection in critically ill patients in Saudi Arabia.

ELIGIBILITY:
Inclusion Criteria:

* adult patients (> 18 years)
* develop invasive candidiasis as per prespecified definitions during ICU stay
* In addition, patients who had invasive candidiasis within 72 hours of ICU admission will be included

Exclusion Criteria:

* Diagnosis of invasive candidiasis (definite or probable) more than 72 hours before ICU admission.
* Diagnosis of invasive candidiasis (definite or probable) within 72 hours of ICU admission, but the admission to ICU for an unrelated reason.
* Readmission to the ICU during the same hospitalization with invasive candidiasis occurring during one of the previous admissions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients (> 18 years) admitted to the ICUs of these centers will be evaluated for the occurrence of Candida infection and followed to discharge or death in ICU. The duration of the study will be 12 months. Also patients who had invasive candidiasis within 72 hours of ICU admission will be included.
Sampling Method: Non-Probability Sample
Enrollment: 162 (Actual)
Dates: Start 2012-08; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hasan Al-Dorzi, MD, Principal Investigator — King Abdulaziz Medical City
Locations (2):
- Saudi Arabia (2):
  - King Abdulaziz Medical City, Riyadh
  - King Fahad Medical City, Riyadh

REFERENCES:
- [Derived] Al-Dorzi HM, Sakkijha H, Khan R, Aldabbagh T, Toledo A, Ntinika P, Al Johani SM, Arabi YM. Invasive Candidiasis in Critically Ill Patients: A Prospective Cohort Study in Two Tertiary Care Centers. J Intensive Care Med. 2020 Jun;35(6):542-553. doi: 10.1177/0885066618767835. Epub 2018 Apr 8. PMID 29628014

RESULTS

PARTICIPANT FLOW:
Groups:
- The Whole Cohort: The whole cohort included one group of patients with invasive candidiasis as per the Inclusion and Exclusion Criteria.
Period: Overall Study
Arm/Group | The Whole Cohort
Started | 162
Completed | 162
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | The Whole Cohort
Number analyzed (Participants) | 162
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.4 (18.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 77
  Male | 85
Region of Enrollment [Number; unit: participants]
  Saudi Arabia | 162

OUTCOME MEASURES:

1. Primary Outcome: Hospital Mortality
Description: For patients staying in the ICU for long periods, hospital mortality will be censored at 180 days after entry into the study.That is patient staying alive in the hospital more than 180 days will be considered alive.
Time Frame: Patients will be followed while in the ICU and the vital status at the time of discharge from the ICU will be noted. The expected stay in the ICU is 10 days on average.
Measure: Count of Participants; unit: Participants
Arm/Group | The Whole Cohort
Number analyzed (Participants) | 162
Participants | 95

2. Secondary Outcome: ICU Mortality
Description: If patients are still alive in the ICU at 180 days after entring the sudy, they will be considered ICU survivors.
Time Frame: patients will be followed until discharge from the hospital and vital status at discharge from the hospital will be noted (expected hospital stay is 5 weeks). Hopsital mortality will be censored at 180 days after entry into the study.
Measure: Count of Participants; unit: Participants
Arm/Group | The Whole Cohort
Number analyzed (Participants) | 162
Participants | 83

3. Secondary Outcome: Duration of Mechanical Ventilation
Description: If multiple intubations in the same admission, then the durations of mechanical ventilation will be added.This will be assessed for up to 180 days of stay in the ICU.
Time Frame: date of extubtation minus date of intubation
Reporting Status: Not Posted

4. Secondary Outcome: Length of Stay in the ICU
Description: Patients will be followed for up to 180 days.Patinets alive in the ICU beyond 180 days of stay will have an ICU length of stay of 180 days.
Time Frame: date of discharge from ICU minus date of admission to ICU
Measure: Mean (Standard Deviation); unit: days
Arm/Group | The Whole Cohort
Number analyzed (Participants) | 162
days | 42.4 (54.2)

5. Secondary Outcome: Length of Stay in the Hospital
Description: Patients will be followed for up to 180 days.Patinets alive in the hospital beyond 180 days of stay will have a hospital length of stay of 180 days.
Time Frame: date of discharge from hospital minus date of admission to hospital
Measure: Mean (Standard Deviation); unit: days
Arm/Group | The Whole Cohort
Number analyzed (Participants) | 162
days | 88.8 (87.2)

ADVERSE EVENTS:
Arm/Group | The Whole Cohort
All-Cause Mortality (participants affected / at risk) | 95/162
Serious Adverse Events (participants affected / at risk) | 0/162
Other Adverse Events (participants affected / at risk) | 0/162

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No